CLINICAL TRIAL: NCT06722976
Title: Digital HEAL (Health and Exercise for Autonomous Longevity)
Brief Title: Digital Health and Exercise for Autonomous Longevity Program
Acronym: DigitalHEAL
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beira Interior (Other)
Responsible Party: Principal Investigator, Ricardo Madeira, PhD Student, University of Beira Interior
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CE-UBI-Pj-2023-064-ID1994; PRT/BD/154440/2022 (Other Grant/Funding Number: FCT-Portuguese Foundation for Science and Technology)
Record Dates: First submitted 2024-11-20; First posted 2024-12-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Mild Cognitive Impairment (MCI); Older People
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- face-to-face (Experimental): The program is organized into three phases: (1) Initial assessment; (2) Multicomponent training sessions; (3) Final assessment.
  1. The initial assessment will consist of physical fitness tests (lasting around 1 hour) and Neuropsychological Assessment tests (lasting around 1.5 hours).
  2. The multicomponent training sessions will last 3 months, twice a week, 50 minutes each session, held in person at the institution.
  3. The final assessment will be the same as the initial assessment (physical fitness tests (about 1 hour) and Neuropsychological Assessment tests (about 1.5 hours).
  Interventions: Other: Multicomponent exercise programs
- Synchronous distance (video call) (Experimental): The program is organized into three phases: (1) Initial assessment; (2) Multicomponent training sessions; (3) Final assessment.
  1. The initial assessment will consist of physical fitness tests (lasting around 1 hour) and Neuropsychological Assessment tests (lasting around 1.5 hours).
  2. The multicomponent training sessions will last 3 months, twice a week, 50 minutes each, carried out by video call.
  3. The final assessment will be the same as the initial assessment (physical fitness tests (about 1 hour) and Neuropsychological Assessment tests (about 1.5 hours).
  Interventions: Other: Multicomponent exercise programs
- Control group (No Intervention): In the control group, the participants take part in the training sessions, and the program is organized into two phases: (1) Initial assessment; (2) Final assessment.
  1. The initial assessment will consist of physical fitness tests (lasting around 1 hour) and Neuropsychological Assessment tests (lasting around 1.5 hours).
  2. The final assessment will be the same as the initial assessment (physical fitness tests (duration approx. 1h) and Neuropsychological Assessment tests (duration approx. 1.5h).
  After completing the assessment, participants will be given the opportunity to do the exercise sessions.

INTERVENTIONS:
Other: Multicomponent exercise programs — The program is organized into three phases: (1) Initial assessment; (2) Multicomponent training sessions; (3) Final assessment.
  1. The initial assessment will consist of physical fitness tests (lasting around 1 hour) and Neuropsychological Assessment tests (lasting around 1.5 hours).
  2. The multicomponent training sessions will last 3 months, twice a week, 50 minutes each session.
  3. The final assessment will be the same as the initial assessment (physical fitness tests (about 1 hour) and Neuropsychological Assessment tests (about 1.5 hours).
  Arms: Synchronous distance (video call); face-to-face

SUMMARY:
Digital HEAL (Health and Exercise for Autonomous Longevity) is a multicomponent training program (combining concurrent training with cognitive stimulation) designed to promote physical fitness and cognitive function in older adults. This program merges a community-based approach with a scientific research project aimed at comparing the effects of in-person and online concurrent training on cognitive function and functional capacity in this population.

The program is structured into three phases: (1) Initial Assessment; (2) Multicomponent Training Sessions; (3) Final Assessment.

1. Initial Assessment The initial assessment will consist of physical fitness tests (approximately 1 hour) and Neuropsychological Evaluation tests (approximately 1.5 hours).
2. Multicomponent Training Sessions The multicomponent training sessions will last for 3 months, with a frequency of two sessions per week, each lasting 50 minutes, conducted in person at the institution.
3. Final Assessment The final assessment will be identical to the initial assessment, comprising physical fitness tests (approximately 1 hour) and Neuropsychological Evaluation tests (approximately 1.5 hours).

Expected Benefits The anticipated benefits for participants include significant improvements in physical fitness, with a particular emphasis on strength, balance, and motor autonomy, which play an essential role in fall prevention. Additionally, cognitive abilities such as orientation, memory, and brain plasticity are expected to improve. The program also aims to promote social interaction, reducing social isolation among older adults. Furthermore, the program will support participants' maintenance within the institution, which helps preserve their routine and address mobility and accessibility limitations. This intervention will also help reduce costs and time for the institution.

Potential Risks The risks associated with participation in the program are similar to those inherent in any physical activity. However, the equipment and environment (floor type, lighting, temperature) are evaluated to ensure suitability for safe exercise at any age. The exercises are supervised by a qualified professional who takes special care to minimize exercise-related risks.

DETAILED DESCRIPTION:
Digital HEAL (Health and Exercise for Autonomous Longevity) is a multicomponent training program (combining concurrent training with cognitive stimulation) designed to promote physical fitness and cognitive function in older adults. This program merges a community-based approach with a scientific research project aimed at comparing the effects of in-person and online concurrent training on cognitive function and functional capacity in this population.

The program is developed and implemented by the Department of Sports Sciences, the Faculty of Health Sciences, and the Department of Psychology and Education of the University of Beira Interior (UBI), in collaboration with the University of Turin. The principal investigator is Ricardo André Alves Bispo Madeira.

The program is structured into three phases: (1) Initial Assessment; (2) Multicomponent Training Sessions; (3) Final Assessment.

1. Initial Assessment The initial assessment will consist of physical fitness tests (approximately 1 hour) and Neuropsychological Evaluation tests (approximately 1.5 hours).
2. Multicomponent Training Sessions The multicomponent training sessions will last for 3 months, with a frequency of two sessions per week, each lasting 50 minutes, conducted in person at the institution.
3. Final Assessment The final assessment will be identical to the initial assessment, comprising physical fitness tests (approximately 1 hour) and Neuropsychological Evaluation tests (approximately 1.5 hours).

Expected Benefits The anticipated benefits for participants include significant improvements in physical fitness, with a particular emphasis on strength, balance, and motor autonomy, which play an essential role in fall prevention. Additionally, cognitive abilities such as orientation, memory, and brain plasticity are expected to improve. The program also aims to promote social interaction, reducing social isolation among older adults. Furthermore, the program will support participants' maintenance within the institution, which helps preserve their routine and address mobility and accessibility limitations. This intervention will also help reduce costs and time for the institution.

Potential Risks The risks associated with participation in the program are similar to those inherent in any physical activity. However, the equipment and environment (floor type, lighting, temperature) are evaluated to ensure suitability for safe exercise at any age. The exercises are supervised by a qualified professional who takes special care to minimize exercise-related risks.

Voluntary Participation and Confidentiality Participation in the program is entirely voluntary, and participants can withdraw at any time without any consequences. Confidentiality is guaranteed, with only the principal investigator, Ricardo André Alves Bispo Madeira, having access to personal data, which will always be coded and not disclosed. The collected data will be used strictly for academic purposes, with no commercial interests. Upon request, individual data can be provided to each participant, improving the assessment of their current condition.

Research Team

The team of researchers involved includes:

Dr. Maria da Assunção Vaz Patto (Associate Professor at the Faculty of Health Sciences, UBI, and researcher at the Health Sciences Research Center - CICS-UBI) Dr. Maria Dulce Leal Esteves (Lecturer in the Department of Sports Sciences and researcher at the Research Center for Sport, Health, and Human Development - CIDESD) Dr. Nuno Filipe Cardoso Pinto (Adjunct Assistant Professor at the Faculty of Health Sciences, UBI, and researcher at CICS-UBI) Ricardo André Alves Bispo Madeira (Ph.D. student in Sports Sciences)

Principal Investigator Signature

By signing this document, I confirm, on behalf of the research team, that I have conveyed all the information contained herein, explained it, and answered all questions and concerns raised by the participant and their family members.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged ≥ 65 years.
* A score of ≥ 3 on the Short Physical Performance Battery (SPPB).
* Willingness to participate in the training programs and collaborate with the research team.

Ability to provide informed consent, either oral or written.

Exclusion Criteria:

* A score of ≤ 3 on the Short Physical Performance Battery (SPPB).
* Presence of severe comorbidities that would negatively impact participation in the training program.
* Presence of color blindness.
* Diagnosis of severe dementia or severe impairment across multiple dimensions of cognition, which would prevent participation in the training program.
* History of surgeries or fractures within the last 6 months.

These criteria ensure that participants are suitable for the program and capable of engaging in the training sessions effectively.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Speed, agility and dynamic balance | 3 months
  The following physical fitness and health parameters will be evaluated:
  6-Minute Walk Test (Distance)
  At the start signal, the subjects were instructed to walk as fast as possible (without running) for 6 minutes. During the test, the supervisor walked slightly behind the participant, avoiding accompanying them side by side so as not to influence the self-selected walking pace.
Speed, agility and dynamic balance | 3 months
  Eight-Foot Up and Go Test (Seconds)
  A chair was placed at the starting point with a cone positioned 8 feet (2.44 m) away. Participants, starting seated with hands on knees, stood up, walked quickly around the cone, and returned to the chair, with timing starting on "go" and stopping when they sat back down.
Strength assessment | 3 months
  The following physical fitness and health parameters will be evaluated:
  Seated Medicine Ball Throw (Meters)
  The seated medicine ball throw test measured upper body strength and power. Participants were seated on a chair, with the trunk against the chair back, holding a 3 kg medicine ball in front of the trunk with both hands. Rotation of the trunk and hips was restricted during the test. Three throws were performed with one-minute rest intervals to prevent fatigue. The distance from the point of release to where the ball contacted the ground was measured using a metric tape. The mean distance of the throws was used for subsequent analysis.
Strength assessment | 3 months
  The following physical fitness and health parameters will be evaluated:
  Arm Curl Test (n. Rep)
  In the arm curl test, participants sat on a chair and were asked to flex the elbow of the strongest arm as many times as possible in 30 seconds while holding a 3 kg dumbbell. Participants were instructed to maintain a normal breathing pattern and keep the elbow at the side of the body throughout the test. A single repetition consisted of complete elbow flexion from maximum extension.
Strength assessment | 3 months
  The following physical fitness and health parameters will be evaluated:
  Handgrip Strength Test (Kg)
  Handgrip strength test, indicative of upper limb muscle function, was measured using an adjustable digital hand dynamometer (Saehan, Model DHD-1, South Korea). Participants were seated with hips, knees, and elbows flexed at 90º, gripping the dynamometer in a neutral forearm position. Three measurements of grip strength were taken for each hand, with a two-minute rest period between attempts. The average of these measurements was used for data analysis.
Strength assessment | 3 months
  The following physical fitness and health parameters will be evaluated:
  Sit-to-Stand Test (n. Rep)
  The sit-stand test was employed to indirectly assess lower limb muscle strength and functionality. Participants used a chair with a 40 cm height and a straight backrest [29]. With arms folded across the chest and plantar support on the floor throughout, participants were instructed to stand up and sit down as many times as possible within 30 seconds. The outcome of this test was determined by counting the number of times the participant successfully completed the sit-stand cycle.
Flexibility assessment | 3 months
  The following physical fitness and health parameters will be evaluated:
  Chair Sit-and-Reach Test (Cm)
  Starting in a seated position, the participant moves their body forwards until they are sitting on the edge of the chair seat. The fold between the top of the leg and the buttocks should be level with the edge of the seat. With one leg bent and the foot fully on the ground, the other leg (the preferred leg) is extended towards the thigh, with the heel on the ground and the foot bent (approx. 90º). The participant should be encouraged to exhale as they flex forwards, avoiding sudden, rapid and strong movements, never reaching the limit of pain.
  With the leg extended (but not hyper-extended), the participant flexes slowly forwards as far as the hip joint (the spine should remain as straight as possible, with the head in the extension of the spine, therefore not flexed), sliding the hands (one over the other, with the fingertips overlapping) along the extended leg, trying to touch the t
Flexibility assessment | 3 months
  The following physical fitness and health parameters will be evaluated:
  Back Scratch Test (Cm)
  In the standing position, the participant places their dominant hand on top of it and reaches as low as possible towards the middle of their back, palm down and fingers extended (elbow pointing upwards). The hand of the other arm is placed underneath and behind, palm facing upwards, trying to reach as far as possible in an attempt to touch (or overlap) the middle fingers of both hands.
Cognitive assessment | 3 months
  The cognitive assessment protocol aims to evaluate multiple dimensions of cognition, including memory, concentration, attention, and executive cognitive functions, as well as their severity. The assessment will include the following validated tests:
  Mini-Mental State Illiterate < 15
  1 to 11 years of schooling < 22 With more than 11 years of schooling < 27
Salivary assessment | 3 months
  Additionally, saliva samples will be analyzed for inflammatory markers such as IL-6 and IL-10, which have been reported in the literature as altered in individuals with dementia
  The assessment of biomarkers was conducted at baseline, after 6 weeks, and post-intervention. To ensure the quality of the samples collected, the experimental collection protocol adhered to strict guidelines. Sampling was consistently performed at the same time (9-11 a.m.) to account for the circadian rhythm of hormones and salivary proteins. The "passive drool" method (unstimulated saliva) was used, where participants sat comfortably, rinsed their mouth with water to remove any residue, and waited 10 minutes before collection began. Saliva was accumulated under the tongue and collected in Falcon tubes. The samples were then transferred to cryotubes and stored at -80 °C.
Salivary assessment | 3 months
  Additionally, saliva samples will be analyzed for inflammatory markers such as TNF-α, which have been reported in the literature as altered in individuals with dementia.
  The assessment of biomarkers was conducted at baseline, after 6 weeks, and post-intervention. To ensure the quality of the samples collected, the experimental collection protocol adhered to strict guidelines. Sampling was consistently performed at the same time (9-11 a.m.) to account for the circadian rhythm of hormones and salivary proteins. The "passive drool" method (unstimulated saliva) was used, where participants sat comfortably, rinsed their mouth with water to remove any residue, and waited 10 minutes before collection began. Saliva was accumulated under the tongue and collected in Falcon tubes. The samples were then transferred to cryotubes and stored at -80 °C.
Body Composition Assessment | 3 months
  Bodyweight (kilogram) BMI The percentage of fat mass was assessed using bioelectrical impedance analysis (BC-BC-613; TANITA, United Kingdom). Body mass index (BMI) was calculated as weight (kg) divided by height squared (m^2). Height measurements were taken using a stadiometer (Cabral, model 14). Participants removed their shoes and stood upright with feet flat on the floor, heels in contact, and their trunk and head positioned together against the stadiometer. The head position was neutral with the chin neither lifted nor tucked. Height measurements were recorded after participants exhaled.
Body Composition Assessment | 3 months
  Free Fat mass (kilogram) Fat mass (%)
  The percentage of fat mass and free fat mass was assessed using bioelectrical impedance analysis (BC-BC-613; TANITA, United Kingdom).
Assessment of memory, concentration, attention and executive cognitive functions | 3 months
  Rey Auditory-Verbal Learning Test scores of ≤10 for more advanced dementia and ≤ 12 for mild/moderate
Assessment of memory, concentration, attention and executive cognitive functions | 3 months
  Verbal Fluency Test (e.g., Units on a Scale) The Verbal Fluency Test is scored based on the total number of words or items generated by the individual.
Quality of Life | 3 months
  Qality of Life PHQ-9 0 to 4: No depression. 5 to 9: Mild depression. 10 to 14: Moderate depression. 15 to 19: Moderately severe depression. 20 to 27: Severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Dulce Esteves, PhD, Study Director — University of Beira Interior
Locations (1):
- Departement of Sports Science, Covilha, Covilhã, Portugal

IPD SHARING:
Plan to Share IPD: Yes
The sharing of individual participant data may be conducted upon request, ensuring that the identification of individuals is always protected to maintain the anonymity of those involved in the research. This approach guarantees the confidentiality and privacy of participants, in accordance with ethical and legal requirements related to data protection.
Time Frame: January 2025 to January 2026
Access Criteria: The data that will support the findings of this study will be available on request from the corresponding author. The request will be analyzed by the research team and the ethics committee that ethically approved the study.

REFERENCES:
- [Background] Hu JP, Guo YH, Wang F, Zhao XP, Zhang QH, Song QH. Exercise improves cognitive function in aging patients. Int J Clin Exp Med. 2014 Oct 15;7(10):3144-9. eCollection 2014. PMID 25419345
- [Background] Janson P, Willeke K, Zaibert L, Budnick A, Berghofer A, Kittel-Schneider S, Heuschmann PU, Zapf A, Wildner M, Stupp C, Keil T. Mortality, Morbidity and Health-Related Outcomes in Informal Caregivers Compared to Non-Caregivers: A Systematic Review. Int J Environ Res Public Health. 2022 May 11;19(10):5864. doi: 10.3390/ijerph19105864. PMID 35627399
- [Background] Tokovska M, Nour MM, Sorensen A, Smaland Goth U. Informal caregivers and psychosocial support: Analysis of European Dementia Policy documents. J Public Health Res. 2021 Sep 27;11(1):2416. doi: 10.4081/jphr.2021.2416. PMID 34579521